

## Institutional Review Board Faculty of Medicine, Chulalongkorn University

The Informed Consent Form

AF 06-07/6.1

page 1/2

Research on Pilot Research Project: Flipping the Paradigm of Parkinson's Disease: A Model of National 'Eat, Move, Sleep' Digital Interventions to Prevent or Slow a Rise of Non-Communicable Diseases in Thailand

| Date | of | Consent | Date | Month | Ye | ar |
|---|---|---|---|---|---|---|
| Mr./M | rs./ľ | Иs | | | | |
| Addre | ess | | | | | |
| Read the details from the information sheet for the participants of the research project attached to the | | | | | | |
| | | | Aı | nd I agree to participate | in the research pr | oject voluntarily. |

I have received a copy of the consent document to participate in the research project that I have signed and the date along with the information documents for the participants of the research project. I was given a detailed explanation by the researcher of the purpose of the research, the duration of the research, the research method, the dangers or symptoms that may arise from the research, as well as the benefits that will arise from the research, and the treatment by other methods. I had enough time and opportunity to ask questions until I understood them well, and the researcher answered the questions with a willingness to hide until I was satisfied.

I acknowledge from the researcher that if any harm arises from such research, I will receive free medical treatment.

I have the right to terminate my participation in the research project at any time. Termination of participation in this research will not affect my treatment or any other rights I may be entitled to. The researcher assures that my personal information will be kept confidential and will only be disclosed with my consent. This must be done for the purpose of verifying the accuracy of the information only. By agreeing to participate in this study, I consent to have my medical history reviewed.

The authors assure that no additional data will be collected. After I have requested to cancel my participation in the research project and want to destroy all documents and/or specimens that can be traced to me.

I understand that I have the right to review or correct my personal information and can revoke the right to use my personal information. The researcher must be informed.

I realized that the data in the research, including my medical information that is not anonymized, goes through processes such as data collection, data collection, and data collection. Recording data in log form and on a computer. Monitoring, analysis, and reporting of data for academic purposes, including future use of medical data, only.



## Institutional Review Board Faculty of Medicine, Chulalongkorn University

The Informed Consent Form

AF 06-07/6.1

page 2/2

I have read the above statement and have understood it well. Willing to participate in research willingly. Therefore, this consent document has been signed.

have read the above statement and have understood it well. Willing to participate in research willingly. Therefore, this consent document has been signed.

| S | igning the Consent |
|------|-------------------------------|
| () | Name of the Consenting Person |
| Date | |

I have explained the objectives of the research, the research method, the dangers, or adverse reactions or risks that may arise from the research, as well as the benefits that will arise from the research, to the participants in the research project named above, who have known and understood it well, and signed a consent document willingly.

| | signed the researcher. |
|------|--------------------------|
| ( | ) Name of the researcher |
| Date | |
| | signed the witness. |
| ( | ) Witness Name Elaborate |
| Data | |